CLINICAL TRIAL: NCT05775913
Title: Development of an Intrauterine Selective Balloon Catheter System for Transcervical Delivery of Selected Agents to the Fallopian Tube
Brief Title: Clinical Evaluation of a Tubal Selective Delivery System
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Jeffrey Jensen, Professor, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: OHSU IRB 24448
Record Dates: First submitted 2022-09-22; First posted 2023-03-20 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Infertility of Tubal Origin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tubal Selective Delivery System (Experimental): The same intervention will be used for all study subjects.
  Interventions: Device: Tubal Selective Delivery System (TSDS)

INTERVENTIONS:
Device: Tubal Selective Delivery System (TSDS) — A novel tubal selective delivery catheter system for selective delivery of administered agents to the fallopian tubes without entry of any portion of the catheter into the tubes.

SUMMARY:
A single center study to evaluate the performance and optimize the design of a novel intrauterine catheter system intended as a nonsignificant risk medical device to aid in evaluating tubal patency as part of the initial diagnostic workup for infertility.

DETAILED DESCRIPTION:
In this study, the investigators will perform transcervical placement of a novel tubal selective delivery catheter system in a controlled clinical setting, using ultrasound imaging to evaluate device performance in a short procedure that will not require sedation or general anesthesia (local anesthesia may be used). The investigator will confirm the position of the device, inflate the balloons, and administer a small volume (10 mL) of an FDA-approved contrast foam. The investigator will then remove the device at the end of the procedure. This study will evaluate performance of the device, ease of use, and patient experience. It will also evaluate the patient experience before, during, and after the procedure. This device is meant to be used to assess tubal patency as part of the initial diagnostic workup for infertility, and use of the device may reduce the need for HSG.

ELIGIBILITY:
Inclusion Criteria:

* Literate in English
* Able to understand and sign an IRB-approved informed consent form
* Willing to complete a pre-procedure questionnaire
* Regular menstrual cycles (24- 38 days)
* Good general health
* Able and willing to comply with all study tests, procedures, and assessment tools
* Uterine sound size between 6 - 10 cm
* Agree to use a non-hormonal method of contraception or avoid vaginal intercourse during the catheter evaluation cycle
* In compliance with cervical cancer screening guidelines per the American Society for Colposcopy and Cervical Pathology (ASCCP) guidelines without evidence of disease.

Alternatively, the subject must have had a colposcopy performed within the appropriate screen time frame, and prior to the study catheter insertion that showed no evidence of dysplasia requiring treatment or further diagnostic procedures or follow-up for at least 6 months

Exclusion Criteria:

* Currently pregnant as confirmed by positive high-sensitivity urine pregnancy test
* Currently using hormonal contraception. Must have at least one natural cycle (two menses) prior to participation if recently discontinued hormonal contraception.
* Currently using an intrauterine device (IUD). Must discontinue at least 30 days prior to Visit 2
* Allergy or hypersensitive to radio-opaque contrast, ExEm foam, both doxycycline and azithromycin (allergy to one not exclusionary if can take the alternative), or lidocaine
* History or physical findings recognized as clinically significant by the investigator, such as symptoms of untreated or recent pelvic infection
* History of involuntary female infertility
* History of gynecologic surgery involving the uterus, fallopian tubes, or ovaries (except single cesarean section)
* History of prior permanent contraception procedure (any technique, abdominal laparoscopic, or hysteroscopic)
* Pelvic exam findings considered clinically-significant by the investigator such as uterine fibroids, pelvic tenderness, or prolapse
* Inability to tolerate placement of a tenaculum and/or uterine sound during screening exam
* Any congenital or acquired uterine anomaly that may complicate study drug placement, such as:

  * Submucosal uterine leiomyoma
  * Asherman's syndromes
  * Pedunculated polyps
  * Bicornuate uterus
  * Didelphys or uterine septa
* Any distortions of the uterine cavity (e.g., fibroids), that, in the opinion of the investigator, are likely to cause issues during insertion, use or removal of the TSDS.
* Known anatomical abnormalities of the cervix such as severe cervical stenosis, prior trachelectomy or extensive conization that, in the opinion of the investigator would prevent cervical dilation and device placement
* Untreated or unresolved acute cervicitis or vaginitis
* Known or suspected human immunodeficiency virus (HIV) infection or clinical AIDS
* Screening transabdominal or transvaginal ultrasound findings with poor imaging quality, or anatomic abnormalities considered clinically important or likely to interfere with assessment of the test device, as assessed by the investigator

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-12 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Clinical performance of catheter during insertion of device | Immediately post-procedure within 30 minutes
  Clinician impression of catheter performance during insertion of device. Performance is categorized as one of three levels: excellent, acceptable, or fail. The number of participants in each category will be reported, with categories defined as:
  Excellent: Clinician can place the insertion tube transcervically without dilation, and advance the obturator to expand the device without the use of imaging guidance.
  Acceptable: Cervical dilation required, but easy to advance the obturator to expand the device without the use of imaging guidance
  Fail: Unable to place the insertion tube
Expansion of arms and dual catheters | During procedure immediately following attempt to position device
  Expansion of arms and dual catheters in the two uterine cornua. Performance is categorized as one of three levels: excellent, acceptable, or fail. The number of participants in each category will be reported, with categories defined as:
  Excellent: Arms extend into bilateral cornua following transcervical insertion after initial expansion. Ultrasound confirms extension but is not needed
  Acceptable: Ultrasound is required to position arms, but expansion is successful after one or two attempts.
  Fail: Clinician is unable to position arms into cornua.
Inflation of dual balloons | During procedure immediate following attempt to inflate balloons
  Inflation of the dual balloons. Performance is categorized as one of three levels: excellent, acceptable, or fail. The number of participants in each category will be reported, with categories defined as:
  Excellent: Inflation of the dual balloons on first attempt by the clinician with no leakage or bad connections. This is confirmed by ultrasound.
  Acceptable: Inflation requires more than one attempt but is ultimately successful.
  Fail: Clinician is unable to inflate balloons due to high pressure or subject pain.
Delivery of saline | During procedure immediate following attempt to administer saline
  Delivery of saline. Performance is categorized as one of three levels: excellent, acceptable, or fail. The number of participants in each category will be reported, with categories defined as:
  Excellent: Successful administration of saline at low pressure (confirmed by ultrasound) with no leakage or bad connections.
  Acceptable: Some leakage of saline, but clinician is able to observe flow in tubes.
  Fail: Clinician unable to administer saline due to high pressure/pain, leakage or bad connections.
Delivery of ExEm foam | During procedure immediate following attempt to administer ExEm foam
  Delivery of ExEm foam. Performance is categorized as one of three levels: excellent, acceptable, or fail. The number of participants in each category will be reported, with categories defined as:
  Excellent: Delivery of foam at low pressure with confirmation of tubal patency via ultrasound and with no leakage or bad connections.
  Acceptable: Some leakage of ExEm in uterine cavity, but clinician is able to observe flow in tubes.
  Fail: Clinician unable to administer ExEm due to high pressure/pain, leakage or bad connections.
Clinician impression of device removal | During procedure immediate following attempt remove device
  Clinician impression of device removal. Performance is categorized as one of three levels: excellent, acceptable, or fail. The number of participants in each category will be reported, with categories defined as:
  Excellent: Clinician can deflate balloons, collapse frame, and withdraw insertion tube without difficulty at the end of procedure without the use of imaging guidance.

SECONDARY OUTCOMES:
Tolerability and ease of use - Provider experience evaluation | Immediately Post-procedure (within 30 minutes)
  The clinician placing the device will evaluate ease of use using a series of 100 mm visual analog scale (anchors: 0 extremely easy; 100 extremely difficult/impossible) to evaluate these questions: Was the device easy to insert transcervically? Was inflation of the balloons easy? Was deliver of saline easy? Was deliver of ExEm foam easy? Was removal easy?
Tolerability and ease of use - Patient experience evaluation | Pre-procedure, during procedure, immediately post-procedure, 15 minutes post-procedure
  Participants will indicate maximum level of pain experienced during study procedures using 100 mm visual analogue scale (VAS) at various time points. We will compare pain with placement, treatment, and removal to several baseline assessments. VAS scales: Baseline expectation of pain, baseline pain immediately following speculum placement, baseline pain immediately prior to placement, pain associated with insertion, pain associated with balloon inflation, pain associated with administration of saline, pain associated with administration of ExEm foam, pain associated with complete device removal, pain 15 minutes after completion of procedure, overall satisfaction with procedure, willingness to recommend procedure to a friend.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Jensen, MD, Principal Investigator — Oregon Health and Science University